CLINICAL TRIAL: NCT05433012
Title: Assessment of the Micro-anatomy of the Menisci and Cartilage in Patients With Presumed Isolated Acute Anterior Cruciate Ligament Injury With Ultrahigh Field MRI at 7T
Brief Title: Assessment Micro-anatomy of the Menisci and Cartilage After Isolated Acute ACL Injury With MRI at 7T
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult Recruiting. Too few patients.
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BASEC-Nr. 2020-02570
Record Dates: First submitted 2022-01-27; First posted 2022-06-27 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Meniscus Lesion; Cartilage Injury; ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isolated Acute Anterior Cruciate Ligament Injury with Ultrahigh Field MRI at 7T (Other)
  Interventions: Device: Ultrahigh Field MRI at 7T

INTERVENTIONS:
Device: Ultrahigh Field MRI at 7T — Assessment of the micro-anatomy of the menisci and cartilage in patients with presumed Isolated Acute Anterior Cruciate Ligament Injury with Ultrahigh Field MRI at 7T

SUMMARY:
Study population The investigator set the sample size to 200 patients.

Primary outcome

* Diagnostic accuracy of ultrahigh field MRI (T7) compared to high field MRI (T3 or less) for detection of meniscal injuries associated with acute ACL injury Secondary outcome
* Influence of 1) Location of injury and 2) meniscal tear pattern (modified WORMS18,19) on the sensitivity of high field MRI compared to ultrahigh field MRI for detection of meniscal tears

DETAILED DESCRIPTION:
However, there is no evidence that ACL reconstruction can actually prevent the development of knee osteoarthritis. However, concomitant meniscal injuries, either at the time of the ACL injury or secondary to the ACL injury, significantly increase the risk of secondary knee osteoarthritis. Therefore, the treatment strategy for ACL injuries is strongly influenced by the presence of concomitant meniscal injuries on initial magnetic resonance imaging (MRI).

To achieve higher spatial resolution and faster image acquisition, there is a clear trend toward higher field strength MRI.

Meniscal injuries repeatedly occur during the course after isolated ACL ruptures, and the question is whether these injuries occurred during the original trauma or as a result of the torn ACL.

Therefore, the primary objective of the current study was to evaluate the potential utility of ultrahigh-field MRI (T7) in detecting occult meniscal tears or cartilage injuries associated with presumed isolated acute ACL injuries compared with high-field MRI (T3 or less). The secondary objective was to evaluate the influence of meniscal tear location and meniscal tear pattern on the sensitivity of high-field MRI compared with ultrahigh-field MRI in detecting meniscal tears. Subsequently, different orthopedic surgeons and radiologists will evaluate the images.

ELIGIBILITY:
Inclusion Criteria:

* Presumed isolated, acute rupture of the anterior cruciate ligament (trauma not older than 4 weeks) diagnosed by high-field MRI (3 Tesla or less) at Balgrist.
* Written informed consent of the study participant
* Age 18 years or older

Exclusion Criteria:

* Previous knee surgery or trauma
* Presence of concomitant meniscal injury on high-field MRI (3 Tesla or less)
* Advanced gonarthrosis (Kellgren-Lawrence score greater than 2).
* Contraindication to the performance of MRI
* Unsigned informed consent
* Inability to follow study procedures (e.g., due to cognitive impairment) or inadequate knowledge of project language
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Frequency of occoult meniscus lesions detected in UHF-MRI | 12 month
  The Menisci are assessed at 6 possible locations in the knee and Meniscal alterations at different locations in the same patient cannot necessarily be considered as independent observations. Therefore, a summary analysis over all 6 possible locations will be conducted to avoid unnecessary multiple testing in separate analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Fucentese, Prof.Dr.med., Study Chair — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland